CLINICAL TRIAL: NCT00836680
Title: Study for the Evaluation of the Efficiency of a Device for the Diagnosis of an Internal Rectal Prolapse, a Pelvic Floor Ptosis and for the Determination of an Internal Hernia Into the Douglas Pouch
Brief Title: Clinical Study for the Evaluation of the Efficiency of a Device for the Diagnosis of an Internal Rectal Prolapse, a Pelvic Floor Ptosis and for the Determination of an Internal Hernia Into the Douglas Pouch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gerhard Pejcl Medizintechnik GmbH (Industry)
Responsible Party: Gerhard Pejcl/Director, Gerhard Pejcl Medizintechnik GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPejcl-230109
Record Dates: First submitted 2009-01-23; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Internal Rectal Prolapse; Pelvic Floor Ptosis; Internal Hernia Into the Douglas Pouch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Colorectal Stent — Diagnosis of an internal rectal prolapse:
  The device will be introduced and placed into the patient via a proctoscopic procedure. After that the doctor can measure and determine the internal rectal prolapse. After the diagnosis results have been received, the device will be removed from the patient via proctoscopic examination. The whole procedure will take approx. 5 minutes.
  An additional X-ray examination procedure with the use of contrast media will be made for the determination of a pelvic floor ptosis and for the determination of an internal hernia into the Douglas pouch.

SUMMARY:
The purpose of this study is to determine if the device is supplying sufficient diagnosis results of an internal rectal prolapse, of a pelvic floor ptosis and for the determination of an interal hernia into the Douglas pouch, as well as to determine the technical success of using the device at the patient.

DETAILED DESCRIPTION:
Existing diagnosis methods are inadequate, inaccurate, complicated or can only made intraoperatively. The new device should enable a fast and easy examination procedure well tolerated by the patients. The diagnosis results, received with the device, should assist in the accurate selection of patients for operations as well as to avoid any unnecessary operations.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* patients with ODS-Symptome-Score according Longo of >7
* existing results about a perceptible and seeable internal rectal prolapse, pelvic floor ptosis and an internal hernia into the Douglas pouch
* patients who correspond to to the ASA 1 - ASA 2 criteria

Exclusion Criteria:

* male patients
* female patients with inflammable or malign diseases of the urogenital tract as well as of the anorectal area and after rectum operation
* female patients with diarrhea
* pregnant patients because of the x-ray examination
* female patients who get anticoagulants
* serious cardiopulmonary disorders
* disorders of the blood coagulation
* female patients who correspond to the ASA 3 to ASA 4 criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Determination if the device will be effective for the diagnosis of an internal rectal prolapse, a pelvic floor ptosis and for the determination of an internal hernia into the Douglas pouch. | 4 months

SECONDARY OUTCOMES:
Determination if the the use of the device will be tolerated by the patient combined with a low level of pain or discomfort. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Abrahamowicz, Dr. med., Principal Investigator
Locations (1):
- St. Elisabeth Hospital, Vienna, Vienna, Austria